CLINICAL TRIAL: NCT02622087
Title: Sex Hormones and Fear Inhibition: a Novel Exploration of Why Women Are so Vulnerable to Anxiety Disorders
Brief Title: The Impact of Sex Hormones on One-session Treatment for Spider Phobia in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of New South Wales (Other)
Responsible Party: Principal Investigator, Bronwyn Margaret Graham, Lecturer and Discovery Early Career Fellow, The University of New South Wales
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MQ13002
Record Dates: First submitted 2015-06-30; First posted 2015-12-04 (Estimated); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Phobia, Specific
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Hormonal contraceptive (Experimental): Women who receive one-session-treatment while they are on the hormonal contraceptive pill
  Interventions: Behavioral: One-Session-Treatment
- Naturally cycling- high estradiol (Experimental): Naturally cycling women who receive one-session-treatment during a period of high estradiol
  Interventions: Behavioral: One-Session-Treatment
- Naturally cycling-low estradiol (Experimental): Naturally cycling women who receive one-session-treatment during a period of low estradiol
  Interventions: Behavioral: One-Session-Treatment

INTERVENTIONS:
Behavioral: One-Session-Treatment — There are a total of five steps, each to be repeated until the participant experiences a reduction of at least 50% in their anxiety. Step 1 is catching a spider with a glass and postcard. Step 2 is touching a spider from behind with the dominant index finger. Step 3 is letting a spider walk on the participant's hands. Step 4 is allowing a spider to walk on the participant's legs and body. Steps 1-4 are repeated with larger spiders, and then the two biggest spiders will walk on the participants' hands simultaneously. Step 5 is using a chopstick to guide a huntsman spider over their gloved hand. Treatment ends when all steps are completed, or if the maximum 3 hour time limit has been reached, or if the participant indicates that they do not want to continue.

SUMMARY:
The purpose of this study is to determine whether levels of sex hormones (including estrogen and progesterone) influence women's response to treatment for Specific Phobia of spiders. It is hypothesised that women will show less relapse of symptoms of spider phobia if they receive treatment during a period of high levels of sex hormones.

DETAILED DESCRIPTION:
Detailed description of the Behavioural Avoidance Test (BAT):

Participants will be asked to stand in front of a closed door. They will be asked by the experimenter to approach the spider as closely as possibly, but they are reminded they can stop at anytime. Participants will then enter a room in which a table will be located approximately 3 meters in front of them. On top of the table will be a glass terrarium containing a fast moving spider (Huntsman - Holconis). These spiders were chosen because they are all low risk (non toxic) and non-aggressive to humans. In addition, these spiders are also commonly found in homes or gardens, thus increasing the ecological validity of our study. Participants will be asked to approach the spider in a stepwise manner (i.e., in 10 steps). Performance will be scored on a 10-point scale that corresponds with the steps taken during the test; the steps are 0 = refuses to enter room, 1 = stops 3m from terrarium, 2 = stops 2m, 3 = stops 1m, 4 = stops close to terrarium, 5 = touches terrarium, 6 = removes lid, 7 = puts hand in terrarium, 8 = touches inside walls and floor of terrarium, 9 = guides spider over hand which is resting on the floor of the terrarium. For steps 7 to 9 the experimenter will relocate the spider to a larger enclosure with a zippered opening that can be arranged so the spider cannot escape the enclosure and the participant will be provided with a long sleeved shirt and a gardening glove. Once the participant has entered the room, the experimenter does not persuade the participant to continue.

Detailed Description of One-Session-Treatment (OST):

There will be three sessions. Session 1 involves the preparation stage, a pre-treatment interview, pre-treatment measures, and OST. During the pre-treatment interview a clinical psychologist will collect information about the participants fear of spiders and provide a rationale for treatment. The participant will then complete pre-treatment measures, including the BAT (to assess pre-treatment levels of avoidance; see detailed protocol above), as well as self-report questionnaires. After completing the pre-treatment measures, participants will then begin OST. This treatment will strictly follow Öst's manual for specific phobias. It will take a maximum of three hours and has been shown to be highly effective in treating specific phobia, including spider phobia. OST involves the use of a maximum of 4 spiders of varying sizes, from 0.5cm to 5cm, housed in glass terrariums. Two spider species will be used: St Andrew's Cross (Argiope) and Huntsman (Holconia immanis). These spiders were chosen because they are all low risk (non toxic) and non-aggressive to humans. In addition, these spiders are also commonly found in homes or gardens, thus increasing the ecological validity of our treatment. There are a total of five steps and at the start of each step, the experimenter will provide instructions and then model the behaviour for the participant. Each step will be repeated until the participant experiences a reduction of at least 50% in their anxiety, as assessed by Subjective Units of Distress ratings (SUDS; 0-100), or rate the conviction in their belief that a catastrophe will occur as 0 (0-100). Steps 1-4 will be completed with the St Andrew's Cross spiders. Step 1 involves teaching the participant how to catch the smallest spider with a glass and postcard (i.e., placing glass upside down over the spider in the terrarium and to slide the postcard underneath). Step 2 involves touching the spider from behind with the dominant index finger. Step 3 involves letting the spider walk on the participant's hands. Step 4 involves allowing the spider to walk on the participant's legs and body. Steps 1-4 are then repeated with larger St Andrew's cross spiders. After completing this, the participant will be encouraged to have the two largest St Andrew's cross spiders walk on their hands simultaneously. Step 5 is provided in the treatment as an extra step and will be completed only if there is time remaining and if the participant gives consent. Step 5 involves encouraging the participant to complete the final step of the BAT using the Huntsman spider (i.e., guiding the spider over their gloved hand). The experiment ends when all steps are completed, or if the maximum 3 hour time limit has been reached, or if the participant indicates that they do not want to continue. After treatment, participants will be checked to ensure they are not feeling any distress and will be accompanied by the experimenter to Healthscope Pathology to provide a blood sample to verify hormone levels.

Session 2, a follow-up session, will occur one-week later, as per Öst's treatment manual. During this session, post-treatment measures will be taken, including structured clinical interview assessment, self-report questionnaires and BAT.

Session 3 will occur 3 months later and will be a long-term follow-up session. Participants will undergo the same measures as in session 2. Participants will be fully debriefed regarding the aims and implications of the experiment. During this process, participants will be asked if they have any questions or concerns, and will be checked to ensure they are not feeling any distress.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-35 with Specific Phobia of Spiders
* Both women who are naturally cycling and women using hormonal contraceptives are eligible to participate

Exclusion Criteria:

* Male
* Certain kinds of comorbid mental illness, including psychosis, bipolar disorder, substance abuse
* Participants with neurological or endocrinological disorders
* In women who are naturally cycling, those who do not have a regular menstrual cycle, are pregnant, or breastfeeding

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in level of approach on the Behavioural Approach Test (BAT) | Pre- treatment, and 1 week and 12 weeks post treatment

SECONDARY OUTCOMES:
Change from baseline in severity of spider phobia on the Spider Phobia Questionnaire | Pre-treatment, and 1 week and 12 weeks post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bronwyn M Graham, PhD, Principal Investigator — University of New South Wales Australia
Locations (1):
- University of New South Wales, Sydney, New South Wales, Australia